CLINICAL TRIAL: NCT00969514
Title: Robotic-assisted Laparoscopic Cystectomy: Our Center's Clinical Experience
Brief Title: Robotic-Assisted Laparoscopic Cystectomy
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Don Bui, Beaumont Hospitals
Other Study IDs: 2009-167
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Cystectomy
Keywords: Robotic cystectomy; Bladder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Robotic cystectomy: Patients undergoing robotic laparoscopic cystectomy at Beaumont Hospital-RO

SUMMARY:
Robotic cystectomy is a relatively new procedure previously described only at university centers. These studies have all been reviews of single surgeon's experiences.

DETAILED DESCRIPTION:
Robotic Cystectomy is a relatively new procedure previously described only at university centers. These studies have all been reviews of single surgeon's experiences. Our objective is to investigate our results from this novel procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robotic cystectomy at Beaumont Hospital

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing robotic cystectomy
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don BUI, MD, Principal Investigator — Beaumont Hospitals-RO
Locations (1):
- Beaumont Hospitals_RO, Royal Oak, Michigan, United States